CLINICAL TRIAL: NCT00005555
Title: Dose Response to Exercise and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Prevention
Other Study IDs: 5099; R01HL058873 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
To determine the minimal dose of physical activity necessary to improve cardiovascular (CV) health by evaluating and aerobically training 500 healthy men and women, 30-65 years of age.

DETAILED DESCRIPTION:
BACKGROUND:

Results from the study will provide important data regarding the dose of exercise required to improve cardiovascular health, as described both by the NIH Consensus Conference on Physical Activity and CV Health and by the recent Report of the Surgeon General. The study was initiated in response to a Program Announcement released in October 1994 on Physical Activity and Cardiopulmonary Health.

DESIGN NARRATIVE:

Subjects were randomized into one of five groups in a 2x2 factorial design plus a usual care control group (n=100 in each of 5 groups). Subjects trained at a moderate (45-55 percent) or high (65-75 percent of maximum heart rate reserve) intensity, and at a frequency of 3-4 or 5-7 days/week (viz., Group 1, 65-75 percent at 5-7 days/week; Group 2, 65-75 percent at 3-4 days/week; Group 3, 45-55 percent at 5-7 days/weekk; Group 4, 45-55 percent at 3-4 days/week; and, Group 5, usual care control). Controls received advice from a physician to increase their physical activity. The subjects in Groups 1-4 participated in an exercise intervention using walking as the mode of training for a total of 24 months. A lifestyle model of physical activity was used, in that subjects could accumulate exercise minutes during the day in 10-minute increments or more continuously (for a total duration of 30 minutes/day), and training was conducted where it was most convenient for the subject (i.e. at home, work or some combination thereof). Tests occurred at baseline (0), 12, and 24 months of the intervention.

The hypothesis was that Groups 1-4 would show a significant reduction in systolic and diastolic blood pressure and an increase in HDL-cholesterol compared to the usual care control group. A second hypothesis was that that there would be significant main effects for both frequency and intensity, with the higher levels of each producing greater improvement on the major outcome variables compared to the lower levels of each dose. The study also planned to determine the minimal dose response to exercise necessary to elicit significant improvement in cardiovascular and behavioral health factors. Finally, the project included examination of the effects of age and level of initial test values on outcome variables to determine if their interactions affected the results of the intervention.

The study also includes assessment of the effect of specific doses of exercise on the reduction in systolic and diastolic blood pressure and increase in HDL-cholesterol (primary outcomes), in addition to changes in levels of physical activity, aerobic fitness (VO2 max), body composition (percent fat and waist-to-hip ratio), triglycerides, and LDL-cholesterol (secondary outcomes). Psychological variables (depression, anxiety, anger, and perceived stress) and health-related quality of life are also evaluated, and the important issue of adherence to exercise is examined with respect to the effect of dose of exercise.

ELIGIBILITY:
No eligibility criteria

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-05; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perri — University of Florida

REFERENCES:
- [Background] Duncan GE, Sydeman SJ, Perri MG, Limacher MC, Martin AD. Can sedentary adults accurately recall the intensity of their physical activity? Prev Med. 2001 Jul;33(1):18-26. doi: 10.1006/pmed.2001.0847. PMID 11482992
- [Background] Perri MG, Anton SD, Durning PE, Ketterson TU, Sydeman SJ, Berlant NE, Kanasky WF Jr, Newton RL Jr, Limacher MC, Martin AD. Adherence to exercise prescriptions: effects of prescribing moderate versus higher levels of intensity and frequency. Health Psychol. 2002 Sep;21(5):452-8. PMID 12211512
- [Background] Duncan GE, Perri MG, Theriaque DW, Hutson AD, Eckel RH, Stacpoole PW. Exercise training, without weight loss, increases insulin sensitivity and postheparin plasma lipase activity in previously sedentary adults. Diabetes Care. 2003 Mar;26(3):557-62. doi: 10.2337/diacare.26.3.557. PMID 12610001
- [Background] Duncan GE, Anton SD, Newton RL Jr, Perri MG. Comparison of perceived health to physiological measures of health in Black and White women. Prev Med. 2003 May;36(5):624-8. doi: 10.1016/s0091-7435(03)00017-3. PMID 12689808
- [Background] Duncan GE, Perri MG, Anton SD, Limacher MC, Martin AD, Lowenthal DT, Arning E, Bottiglieri T, Stacpoole PW. Effects of exercise on emerging and traditional cardiovascular risk factors. Prev Med. 2004 Nov;39(5):894-902. doi: 10.1016/j.ypmed.2004.03.012. PMID 15475021